# A Phase 3 Multicenter Study of the Long-term Safety and Tolerability of ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder in Adults who Have an Inadequate Response to Antidepressant Therapy (the FORWARD-2 Study)

**Unique Protocol ID:** ALK5461-208

NCT Number: NCT02141399

**EudraCT Number:** 2014-000380-41

**Date of Statistical Analysis** 

Plan: 15 September 2017



# STATISTICAL ANALYSIS PLAN PHASE III

#### ALK5461-208

Study Title: A Phase 3 Multicenter Study of the Long-term Safety and

Tolerability of ALKS 5461 for the Adjunctive Treatment of

Major Depressive Disorder in Adults who Have an Inadequate Response to Antidepressant Therapy (the

FORWARD-2 Study)

Document Status: Final

Document Date: 15 September 2017

Based on: Study protocol amendment 3 (dated 03 March 2016)

Study protocol amendment 2 (dated 12 May 2015)

Study protocol amendment 1 (dated 17 April 2014)

Original study protocol (dated 16 December 2013)

Sponsor: Alkermes, Inc.

852 Winter Street Waltham, MA 02451

USA

#### **CONFIDENTIAL**

Information and data in this document contain trade secrets and privileged or confidential information, which is the property of Alkermes, Inc. No person is authorized to make it public without the written permission of Alkermes, Inc. These restrictions or disclosures will apply equally to all future information supplied to you that is indicated as privileged or confidential. This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

# TABLE OF CONTENTS

| LIST OF | ABBREVIATIONS | 5 |
|----------|---------------------------------------------------------|----|
| 1. | INTRODUCTION | 7 |
| 1.1. | Study Objectives | 7 |
| 1.2. | Summary of the Study Design and Schedule of Assessments | 7 |
| 1.3. | Criteria for Evaluation | 9 |
| 2. | SAMPLE SIZE AND STATISTICAL POWER CONSIDERATION | 10 |
| 3. | DATA ANALYSIS | 10 |
| 3.1. | General Statistical Methodology | 10 |
| 3.2. | Study Population | 10 |
| 3.2.1. | Definitions of Analysis Populations (Analysis Sets) | 10 |
| 3.2.2. | Disposition | 13 |
| 3.2.3. | Protocol Deviations | 13 |
| 3.3. | Demographics and Baseline Characteristics | 14 |
| 3.4. | Prior and Concomitant Medications | 14 |
| 3.5. | Treatment Adherence Rate and Extent of Exposure | 15 |
| 3.6. | Efficacy Analysis | 16 |
| 3.6.1. | General Considerations | 16 |
| 3.6.1.1. | Pooling of Centers | 16 |
| 3.6.1.2. | Multiple Comparisons/Multiplicity | 16 |
| 3.6.1.3. | Examination of Subgroups | 16 |
| 3.6.2. | Efficacy Analysis | 16 |
| 3.6.2.1. | Montgomery-Asberg Depression Rating Scale (MADRS) | 16 |
| 3.6.2.2. | Hamilton Rating Scale for Anxiety (HAM-A) | 17 |
| 3.6.2.3. | Clinical Global Impression – Severity (CGI-S). | 17 |
| 3.7. | Safety Analysis | 18 |
| 3.7.1. | General Considerations | 18 |
| 3.7.2. | Adverse Events | 18 |
| 3.7.3. | Adverse Events of Special Interest | 20 |
| 3.7.4. | Clinical Laboratory Parameters | 21 |
| 3.7.4.1. | Descriptive Analysis of Laboratory Parameters | 21 |
| 3.7.4.2. | Outlier Analyses of Laboratory Parameters | 22 |

| 3.7.4.3. | Hepatic Effects | 25 |
|---|---|---|
| 3.7.5. | Vital Signs | 26 |
| 3.7.6. | Electrocardiograms | 27 |
| 3.7.7. | Columbia Suicide Severity Rating Scale (C-SSRS) | 28 |
| 3.7.8. | Clinical Opiate Withdrawal Scale (COWS) Scores | 31 |
| 4. | INTERIM ANALYSES | 32 |
| 5. | CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL | 32 |
| 6. | DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA | 32 |
| 6.1. | Analysis Visit Windows | 32 |
| 6.2. | Efficacy Data Handling | 32 |
| 6.3. | Handling of Partial Dates of Prior and Concomitant Medications | 33 |
| 7. | GENERAL STATISTICAL METHODOLOGY | 33 |
| 7.1. | Statistical Conventions | 33 |
| 7.2. | Reporting Precision | 33 |
| 8. | PROGRAMMING SPECIFICATIONS | 34 |
| 9. | MOCK TABLES, LISTINGS AND FIGURES (TLFS) | 34 |
| 10. | REFERENCES | 34 |
| APPEND | IX 1. AESI – ABUSE POTENTIAL | 35 |
| APPEND | IX 2. AESI – DEPENDENCE | 37 |
| APPEND | IX 3. AESI – WITHDRAWAL | 38 |
| APPEND | IX 4. AESI – SUICIDAL IDEATION AND BEHAVIOR | 40 |
| APPEND | IX 5. AESI – HYPOMANIA/MANIA | 41 |
| APPEND | IX 6. AESI – CNS DEPRESSION AND SEDATION | 42 |
| APPEND | IX 7. AESI – RESPIRATORY DEPRESSION | 43 |
| APPEND | IX 8. AESI – ORTHOSTASIS HYPOTENSION | 44 |
| APPEND | IX 9. AESI – HYPERSENSITIVITY | 45 |
| APPEND | IX 10. AESI – SLOWING OF VENTRICULAR REPOLARIZATION | 53 |
| APPEND | IX 11. AESI – HEPATIC EFFECTS | 54 |
| APPEND | IX 12. AESI – SEXUAL DYSFUNCTION | 57 |

# LIST OF TABLES

| Table 1: | Schedule of Safety Assessments. | 9 |
|---|---|---|
| Table 2: | Baseline and Study Period for Safety Endpoints | 12 |
| Table 3: | Definitions to Define Study Drug Cumulative Exposure | 15 |
| Table 4: | Potentially Clinically Significant Abnormal Laboratory Values | 23 |
| Table 5: | Shift Criteria and Denominator for Alanine Aminotransferase (ALT) | 25 |
| Table 6: | Shift Criteria and Denominator for Aspartate Aminotransferase (AST) | 26 |
| Table 7: | Shift Criteria and Denominator for Total Bilirubin (TBILI) | 26 |
| Table 8: | Potentially Clinically Significant Abnormal Vital Sign Values | 27 |
| Table 9: | Potentially Clinically Significant Abnormal ECG Values | 28 |
| Table 10: | C-SSRS Summary Categories for Analysis | 29 |
| Table 11: | Treatment Emergent Suicide-related Events for Analysis | 30 |
| Table 12: | Degree of Precision. | 33 |
| | LIST OF FIGURES | |
| Figure 1: | Study Design Schematic | 8 |

# LIST OF ABBREVIATIONS

The following abbreviations are used in the statistical analysis plan.

| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| ADT | Antidepressant Therapy |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| BDZ | Benzodiazapine |
| BMI | Body Mass Index |
| BUP | Buprenorphine |
| CGI-S | Clinical Global Impression - Severity |
| CI | Confidence Interval |
| CNS | Central Nervous System |
| COWS | Clinical Opiate Withdrawal Scale |
| CRF | Case Report Form |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DILI | Drug Induced Liver Injury |
| ECG | Electrocardiogram |
| eDISH | Evaluation of Drug-induced Serious Hepatotoxicity |
| EOT | End of Treatment |
| ET | Early Termination |
| FAS | Full Analysis Set |
| HAM-A | Hamilton Rating Scale for Anxiety |
| LLRR | Lower Limit of Reference Range |
| MADRS | Montgomery-Asberg Depression Rating Scale |
| MAOI | Moclobemide |
| MDD | Major Depressive Disorder |
| MDE | Major Depressive Episode |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NDA | New Drug Application |
| PCS | Potentially Clinically Significant |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------------|
| PDEAE | Post-discontinuation Emergent Adverse Event |
| PLI | Prospective Lead-in |
| PT | Preferred Term |
| QTcF | QTcF – Fridericia's Correction Formula |
| SAE | Serious Adverse Event |
| SAM | Samidorphan |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SE | Standard Error |
| SNRI | Serotonin-norepinephrine Reuptake Inhibitor |
| SOC | System Organ Class |
| SSRI | Selective Serotonin Reuptake Inhibitor |
| TBILI | Total Bilirubin |
| TCA | Tricyclic Antidepressant |
| TEAE | Treatment Emergent Adverse Events |
| ULRR | Upper Limit of Reference Range |
| VS | Vital Sign |
| WHO-ATC | World Health Organization Anatomical Therapeutic Chemical |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical methods and data presentation to be used for analyzing and reporting efficacy and safety data for study ALK5461-208 for the adjunctive treatment of Major Depressive Disorder (MDD) at study completion. This document has been prepared based on Alkermes ALK5461-208 study protocol amendment 3 (dated 03 March 2016) [1].

# 1.1. Study Objectives

The objective of this study is to assess the long-term safety and tolerability of ALKS 5461 for use as an adjunctive therapy to antidepressants for the treatment of MDD.

### 1.2. Summary of the Study Design and Schedule of Assessments

This is a Phase 3, multicenter, multinational, study to evaluate the long-term safety and tolerability, and to explore treatment effect of 52 weeks of ALKS 5461 administration for use as an adjunctive therapy to antidepressants (ADT) for the treatment of MDD in subjects who have had 1 or 2 inadequate response to an approved ADT in the current MDE.

ALKS 5461 was studied at a dose of 2 mg buprenorphine (BUP):2 mg samidorphan (SAM). Note that ALKS 5461 dose levels are referred to as doses of BUP/SAM expressed as weight in mg (eg, a 2 mg BUP:2 mg SAM dose is expressed as ALKS 5461 2/2).

All subjects in the study had been treated with an adequate dose of an approved ADT for at least 8 weeks, at a stable dose over the last 4 weeks prior to study entry.

Subjects will enter into the study in one of three ways, based on their prior experience with an ALKS 5461 study:

- 1. New Subjects: those who have not participated in a prior study of ALKS 5461 within 2 years.
- 2. <u>Continuing Subjects</u>: those who have completed the treatment period of study ALK5461-205, ALK5461-206, ALK5461-207, or ALK5461-210 within the past 10 days. Since some of these antecedent studies were randomized placebo-controlled studies, these subjects may or may not have received ALKS 5461 in the prior study.
- 3. <u>Lead-in Subjects</u>: those who participated in study ALK5461-205, ALK5461-206, or ALK5461-207 within the past 10 days, and met the criteria for response to ADT during the prospective lead-in (PLI) period of that antecedent study, but did not meet the criteria for remission. These subjects were not eligible for entry into the double-blind treatment period in the antecedent and received neither placebo nor ALKS 5461 in the antecedent study.

All New Subjects will be initially evaluated for eligibility at screening (Visit 1), to occur up to 28 days prior to Visit 2.

For Continuing Subjects and Lead-in Subjects, Visit 2 will be the first visit of this study and there will not be a separate screening visit. Identical assessments taken at the subject's last visit

of the antecedent study do not need to be repeated at Visit 2 of this study unless more than 10 days elapses between these visits.

At Visit 2, all eligible, consenting subjects will begin the treatment period. Subjects entering the study already receiving ALKS 5461 will not require titration; all other subjects will require a 1-week ALKS 5461 titration period. Depending on the antecedent study, the titration may be blinded per blinding schemes as described in the protocol. From Week 2 to 52, all participating subjects will take ALKS 5461 2/2 and an approved ADT, with allowable ALKS 5461 dose adjustments for tolerability as described in the protocol.

During the 52-week treatment period, subjects will return to the clinic for periodic scheduled visits (Visits 2-14) at which safety, tolerability, and treatment effect over time will be assessed.

A 4-week safety follow-up period will occur following the ALKS 5461 treatment period. During the 4-week follow-up period, there are a total of 4 clinic visits (Visits 15-18), as well as 7 safety assessments by phone. Please refer to the protocol for a detailed schedule of assessments. A brief schematic of study design is provided in Figure 1. A summary of the schedule of safety assessments is presented in Table 1.

Figure 1: Study Design Schematic



Abbreviations: EOS=end of study; EOT=end of treatment; ET=early termination; PLI=prospective lead-in; V=visit

**Table 1:** Schedule of Safety Assessments

| Study<br>Number | Dosing<br>Schedule<br>(Days) | Vital<br>Signs <sup>a</sup> | Clinical<br>Laboratory<br>Testing <sup>b</sup> | 12-Lead<br>ECG | C-SSRS <sup>d</sup> | COWS <sup>e</sup> | AEs |
|---|---|---|---|---|---|---|---|
| ALK5461-<br>208 | Treatment:<br>1-365 (1<br>year)<br>Titration:<br>1-7 (1<br>week)<br>Safety<br>Follow<br>Up: 366-<br>393 (1<br>month) | Screening,<br>Days 1°, 8,<br>15, 29, 43,<br>57, 99, 141,<br>183, 225,<br>267, 309,<br>365, 366,<br>372, 379,<br>393 | Screening,<br>Days 1°, 8,<br>99, 183,<br>267, 365,<br>393 | Screening,<br>Days 1°,<br>8, 183,<br>365, 393 | Screening,<br>Days 1°, 8,<br>15, 29, 43,<br>57, 99, 141,<br>183, 225,<br>267, 309,<br>365, 366,<br>372, 379,<br>393 | Days<br>365,<br>366,<br>372,<br>379,<br>393 <sup>e</sup> | Throughout |

Abbreviations: ECG=electrocardiogram; C-SSRS=Columbia-Suicide Severity Rating Scale; COWS=Clinical Opiate Withdrawal Scale; AEs=Adverse Events

#### 1.3. Criteria for Evaluation

#### Safety and Tolerability:

The following assessments will be collected to measure safety and tolerability throughout the study:

- Adverse events (AEs)
- Vital signs (VS)
- Weight
- Clinical laboratory parameters (chemistry, hematology, and urinalysis)
- Electrocardiogram (ECG) parameters
- Columbia Suicide Severity Rating Scale (C-SSRS)
- Clinical Opiate Withdrawal Scale (COWS)

#### **Efficacy:**

The following assessments will be collected to measure treatment effect throughout the study:

- Montgomery-Asberg Depression Rating Scale (MADRS)
- Hamilton Rating Scale for Anxiety (HAM-A)
- Clinical Global Impression Severity (CGI-S)

<sup>&</sup>lt;sup>a</sup> Vital signs included weight, oral temperature, supine respiratory rate, blood pressure, and heart rate.

<sup>&</sup>lt;sup>b</sup> Chemistry, hematology, and urinalysis.

<sup>&</sup>lt;sup>c</sup> Conducted predose.

d At screening the "Baseline" version of the C-SSRS was administered and at all other visits the "Since Last Visit" version was administered.

<sup>&</sup>lt;sup>e</sup> COWS was administered by a medical professional.

#### 2. SAMPLE SIZE AND STATISTICAL POWER CONSIDERATION

Approximately 1,500 subjects will be enrolled in order to achieve at least 100 subjects with 12 months and 300 subjects with 6 months of exposure to ALKS 5461. Subjects will enter from four feeder studies or enter de novo. The antecedent studies included ALK5461-205, ALK5461-206, ALK5461-207, and ALK5461-210.

#### 3. DATA ANALYSIS

#### 3.1. General Statistical Methodology

The safety and efficacy endpoints will be summarized by prior ALKS 5461 exposure: no prior exposure to ALKS 5461 and prior exposure to ALKS 5461, as well as overall.

<u>Subjects with no prior exposure to ALKS 5461</u> come from three sources: De Novo (i.e., New Subjects), PLI Failures (i.e., antecedent study Prospective Lead-in Subjects Failures) and Placebo (i.e., those who did not receive any active treatment in an antecedent study).

<u>Prior exposure to ALKS 5461 subjects</u> include Continuing Subjects who received active treatment (doses ALKS 5461 0.5/0.5, ALKS 5461 1/1, or ALKS 5461 2/2) in an antecedent study. Subjects with prior exposure are designated as such independent of the duration of exposure in the antecedent trial.

In general, summary statistics (n, mean, standard deviation [SD], median, minimum, and maximum for continuous variables, and number and percentage of subjects in each category for categorical variables) based on observed data will be provided by prior ALKS 5461 exposure and overall. Measurements collected from unscheduled visits or repeated assessments will not be included in the by-visit summary tables or figures, but will be included in categorical outlier analyses of post-baseline values and subject listings.

In general, only data collected during the ALK5461-208 study will be summarized even though the baseline may come from an antecedent study.

Last assessment during treatment period, defined as the last non-missing value from scheduled post-baseline visit during the treatment period (i.e., from Visit 2 to Visit 14, inclusive), will be included in the by-visit summary tables for both efficacy and safety endpoints as appropriate.

Source data for the summary tables will be presented as subject data listings. Please refer to Section 6.1 on the handling of data collected at an early termination visit.

# 3.2. Study Population

#### 3.2.1. Definitions of Analysis Populations (Analysis Sets)

<u>Safety Population</u> consists of all subjects who receive at least 1 dose of study drug in the ALK5461-208 study.

An AE will be considered as a treatment emergent adverse event (TEAE) if it starts or worsens (if present at baseline) on or after the baseline during treatment period. An AE will be

considered as a post-discontinuation emergent adverse events (PDEAE) if it starts or worsens after the last dose date plus 1 day.

<u>Post-discontinuation Safety Population</u> consists of subjects in the Safety Population who have at least 1 post-discontinuation measurement. There will be two Post-discontinuation Safety Populations, one is used to analyze PDEAE, and the other is to analyze COWS, grouped by whether having had exposure to study drug in a prior controlled trial or had no prior exposure.

<u>Post-discontinuation Safety Population for PDEAE</u> consists of subjects who received at least 1 dose of study drug, and met one of the following criteria:

- Subjects who entered the Post-discontinuation Period and had a Post-discontinuation Visit
- Subjects who did not enter the Post-discontinuation Period, but had at least 1 PDEAE reported
- Subjects who died after either completing the treatment or having an Early Termination (ET) Visit

<u>Post-discontinuation Safety Population for COWS</u> consists of subjects who received at least 1 dose of study drug, had an adequate COWS baseline (defined as end of treatment [EOT] COWS assessment) and had at least 1 post-EOT COWS assessment, where an adequate EOT COWS is defined as having been performed within (≤) 2 days of last dose of study drug.

<u>Full Analysis Set (FAS)</u> consists of subjects in the Safety Population who have at least 1 post-baseline complete MADRS assessment.

The baseline for efficacy endpoints is defined as the last non-missing observation on or before the date of baseline visit (Visit 2) of ALKS 5461-208 study for subjects who are new to ALKS 5461 (ie, De Novo, PLI Failures, and Continuing Subjects who received placebo in antecedent study); or the last non-missing observation on or before the first dose of ALKS 5461 in antecedent study for Continuing Subjects who received any dose of ALKS 5461 (i.e., ALKS 5461 0.5/0.5, ALKS 5461 1/1, or ALKS 5461 2/2) in antecedent study.

The baseline and study period are defined in Table 2 for each safety endpoint. Visit 2 is the first scheduled visit during treatment period and Visit 14 is the last scheduled visit including ET visit during treatment. Please refer to Protocol for detailed schedule of assessments.

 Table 2:
 Baseline and Study Period for Safety Endpoints

| Safety Endpoint | Population | Study Period and Baseline |
|---|---|---|
| AE | Safety Population | For AEs, treatment period will include the interval between the date of Visit 2 and the last dose date plus 1 day, inclusive. |
| | | For new subjects, the baseline for TEAEs is defined as all AE data collected prior to Visit 2 in Study ALK5461-208. For all other subjects, Visit 2 will be their first visit of this study, so all the AEs occurred or worsened after Visit 2 during treatment period are considered as TEAE. |
| Lab, VS , ECG<br>and C-SSRS | Safety Population | For safety endpoints lab, VS, ECG and C-SSRS, the treatment period will include assessments collected at the Visit 2 baseline visit and all post-baseline visits throughout the entire treatment period starting from Visit 2 to the last assessment visit date. |
| | | The baseline for these safety endpoints is defined as the last non-missing value on or before the date of Visit 2. |
| PDEAE | Post-discontinuation<br>Safety Population<br>for PDEAE | For PDEAEs, the Post-discontinuation Safety Period will be defined as the interval starting from the last dose date plus 2 days to the end of study date. The baseline for PDEAEs is defined as all data collected prior to last dose date plus 2 days. |
| Safety Population covers the value | | For COWS, Post-discontinuation Safety Period covers the values collected from the EOT visit (Visit 14) through the post-discontinuation visits. |
| | | The post-discontinuation baseline for COWS is defined as EOT COWS assessment (Visit 14), and an adequate post-discontinuation baseline is defined as EOT COWS having been performed within (≤) 2 days of last dose of study drug. |

#### 3.2.2. Disposition

Subject disposition will be summarized for all subjects and for subjects categorized as having prior ALKS 5461 exposure and no prior ALKS 5461 exposure. Subjects with no prior ALKS 5461 exposure will be further summarized by the following sub-categories: De Novo (i.e., New Subjects), PLI Failures (i.e., Lead-in Subjects), and Placebo (i.e., Continuing subjects who received only placebo in the antecendent study). The number and percentage of subjects will be summarized for the following:

- Subjects who enrolled in the study
- Subjects in the Safety Population
- Subjects in the FAS population
- Subject who completed treatment (as indicated on the case report form, CRF)
- Subjects who completed the study (as indicated on the CRF)
- Subjects who discontinued from the study

For subjects who prematurely discontinue from the study, the reasons for discontinuation as recorded on the disposition CRF will be presented. Percentage will be calculated based on Safety Population. Disposition for those subjects who had a down-titratration from the ALKS 5461 2/2 mg dose will be summarized similarly.

A listing of disposition will be provided for all subjects.

Additional analysis will include analysis of time to treatment discontinuation for subjects who discontinue from the study. Time to treatment discontinuation will be summarized for those with study discontinuation due to any cause and due to AE as indicated on the disposition CRF. For those subjects who discontinued due to AE or due to any other reason, time to discontinuation will be calculated from the date of the first dose of ALKS 5461 in the ALK5461-208 study (Visit 2), to the EOT visit date. In analysis of time to treatment discontinuation due to AE, subjects who discontinue for other reasons will be censored by day of EOT. The distribution of time to treatment discontinuation will be estimated and graphically displayed by prior ALKS 5461 experience and overall using Kaplan-Meier methods. Time to treatment discontinuation will also be summarized by descriptive statistics.

#### 3.2.3. Protocol Deviations

Subjects with major protocol deviations will be summarized by prior ALKS 5461 exposure and overall along with supportive listings for each of the following categories:

- Did not meet the inclusion / exclusion criteria
- Received prohibited medications
- Lack of adherence with study medication, as defined by subjects taking less than 70% of the protocol specified amount of study medication
- Dosing error
- Other major protocol deviation

#### 3.3. Demographics and Baseline Characteristics

For New Subjects only, demographic and baseline characteristics data (including MDD history) will be collected at screening visit. For Continuing Subjects and Lead-in Subjects, these data will be carried over from information recorded in the antecedent ALKS 5461 study in which they participated.

Demographics and baseline characteristics (age, gender, primary race, ethnicity, region (United States [US], non-US), duration of current MDE, ADT Class for current MDE, number of inadequate responses to ADT in the current MDE, lifetime number of MDEs, lifetime number of antidepressants, benzodiazepines (BDZ) use, opioid use, H1 antagonist use, height, weight, body mass index [BMI]) will be summarized by prior exposure to ALKS 5461, no prior exposure to ALKS 5461, and overall for the Safety Population. For no prior exposure to ALKS 5461, the group is divided further into 3 subgroups of De Novo, PLI Failures, and Placebo, as well as overall. Categories for missing data will be provided as necessary.

Baseline characteristics for efficacy measurments (MADRS-10 score, MADRS-6 score, HAM-A total score, CGI-S score and HAM-D total score) will be summarized by prior exposure to ALKS 5461, no prior exposure to ALKS 5461, and overall for the FAS Population. For no prior exposure to ALKS 5461, the group is divided further into three subgroups of De Novo, PLI Failures, and Placebo, as well as overall. The baseline for efficacy measurements is defined as the last non-missing value on or before the date of initiation of ALKS 5461 at any dose.

Medical and psychiatric history will be summarized using the number of observations and percentage of subjects reporting each category by prior ALKS 5461 exposure and overall for the Safety Population.

Demographic and baseline listings will be provided for all subjects.

#### 3.4. Prior and Concomitant Medications

Prior medications are defined as medications started prior to the first dose of study drug. Concomitant medications are defined as medications taken during the period between the first dose date and the last dose date of study drug, inclusive. All medications as documented by the investigator will be coded using the World Health Organization Anatomical Therapeutic Chemical (WHO-ATC) drug dictionary version June 2016.

Prior medications and concomitant medications will be summarized by ATC code and Preferred Term, by Preferred Term, and by prior ALKS 5461 exposure and overall for the Safety Population. For the summary tables, if a subject has taken a prior or concomitant medication more than once, the subject will be counted only once for the medication.

In addition, the prior and concomitant ADTs by ADT class (selective serotonin reuptake inhibitor [SSRI], serotonin-norepinephrine reuptake inhibitor [SNRI], Tricyclic Antidepressant [TCA], Moclobemide [MAOI] and other) and Preferred Term will be summarized similarly.

Summary tables for benzodiazepines use, opioid use, and sedating H1 antagonist use (prior medication / concomitant medication) by Preferred Term and by prior ALKS 5461 exposure and overall for the Safety Population will be produced, respectively.

A list of subjects taking ADTs, Benzodiazepines (BDZ) and BDZ-like drugs, Opioids, and sedating H1 antagonists will be provided.

#### 3.5. Treatment Adherence Rate and Extent of Exposure

Treatment adherence to the daily dosing schedule of study drug is measured as the rate of actual compared to intended number of doses to be taken during the ALK5461-208 study. Percentage of treatment adherence will be calculated during 52-week treatment period for the Safety Population as follows:

 $\frac{\text{Total tablets taken}}{\text{Total tablets subject should have taken from the first dose date to the last dose date, inclusive}}$ 

Duration of exposure to study drug is defined as the number of days from the first dose date of study drug taken to the date of the last dose taken during the ALK5461-208 study, inclusive.

Treatment adherence and exposure of study drug will be summarized by prior ALKS 5461 exposure and overall for the Safety Population.

Treatment adherence will be summarized as a continuous measure using descriptive statistics (number of subjects, mean, SD, median, minimum, and maximum) and as a categorical measure using the number and percentage of subjects in each adherence rate category (rounded to the whole number): <70%;  $\ge70\%$  to 80%; >80% to 90%; >90% to 100%; >100% to 110%; >110% to 119%; and  $\ge120\%$ .

The number of subjects exposed to study drug and the average days of treatment will be summarized as a continuous measure using descriptive statistics (number of subjects, mean, SD, median, minimum, and maximum).

The exposure to ADT will be summarized by ADT class (SSRI, SNRI, TCA, MAOI and other) and Preferred Term (ADT name) using descriptive statistics in a similar fashion. In addition, descriptive statistics of mean daily dose of ADT will be summarized by ADT class and Preferred Term.

The descending cumulative exposure of study drug will be categorized as  $\ge 1$  day,  $\ge 1$  month,  $\ge 3$  months,  $\ge 6$  months,  $\ge 9$  months and  $\ge 12$  months, and will be summarized as a categorical measure using the number and percentage of subjects in each category.

The definitions in Table 3 will be used to define cumulative exposure.

**Table 3:** Definitions to Define Study Drug Cumulative Exposure

| | Definition | <b>Programming Derivation</b> |
|-----------------|---------------------------|--------------------------------|
| ≥ 1 day | ≥ 1 day | |
| ≥ 1 month | ≥ 23 days (3 weeks) | $\geq$ (365.25/12)-7 days |
| $\geq$ 3 months | $\geq$ 84 days (12 weeks) | $\geq$ [(365.25/12)x3]-7 days |
| ≥ 6 months | ≥ 169 days (24 weeks) | $\geq$ [(365.25/12)x6]-14 days |
| ≥ 9 months | ≥ 260 days (37 weeks) | $\geq$ [(365.25/12)x9]-14 days |
| ≥ 12 months | ≥ 351 days (50 weeks) | ≥ 365.25 -14 days |

#### 3.6. Efficacy Analysis

#### 3.6.1. General Considerations

All efficacy analyses will be based on the FAS. Descriptive statistics will be summarized by prior ALKS 5461 exposure and overall based on observed data.

#### 3.6.1.1. Pooling of Centers

No plan to pool study centers.

#### 3.6.1.2. Multiple Comparisons/Multiplicity

Not applicable.

#### 3.6.1.3. Examination of Subgroups

No subgroup analysis for efficacy is planned.

#### 3.6.2. Efficacy Analysis

#### 3.6.2.1. Montgomery-Asberg Depression Rating Scale (MADRS)

The MADRS measures the severity of depressive symptoms and consists of 10 items. The MADRS-10 is the sum of all 10 items and ranges from 0 to 60. The MADRS-6 is the sum of the following 6 items: item 1 reported sadness; item 2 apparent sadness; item 3 inner tension; item 7 lassitude; item 8 inability to feel; and item 9 pessimistic thoughts and ranges from 0 to 36. Section 6.2 describes the handling of MADRS-10 if any of the items of the MADRS is missing.

The following endpoints will be assessed:

- Change from baseline in MADRS-10 and MADRS-6 score
- Proportion of subjects demonstrating MADRS treatment response, defined as a ≥50% reduction in MADRS-10 from baseline
- Proportion of subjects achieving remission, defined as a MADRS-10 of  $\leq$ 10

Descriptive summary statistics of baseline MADRS-10 and MADRS-6 score and change from baseline at each visit including the last assessment during treatment period will be provided by prior ALKS 5461 exposure and overall based on observed data. In addition, the figures of MADRS-10 and MADRS-6 score (including standard error), mean change from baseline (including standard error) over time including the last assessment during treatment period will be provided by prior ALKS 5461 exposure and overall based on observed data.

The responder and remission endpoints are derived based on the observed MADRS-10. The number and percentage of subjects demonstrating MADRS-10 treatment response and remission by visit including the last assessment during treatment period will be provided based on FAS. The figures of MADRS-10 responder rate and MADRS-10 remission rate over time including the last assessment during treatment period will be provided by prior ALKS 5461 exposure and overall.

The individual MADRS item scores will not be summarized but will be included in the subject listing.

#### **3.6.2.2.** Hamilton Rating Scale for Anxiety (HAM-A)

The HAM-A is a clinician-administered 14-item scale developed to measure the severity of anxiety symptoms. The HAM-A total score is the sum of all 14 items and ranges from 0 to 56. Section 6.2 describes the handling of total score if any of the items of the HAM-A is missing.

The following endpoints will be assessed

- Change from baseline in HAM-A total score
- Change from baseline in HAM-A psychic subscale, where the psychic subscale is the sum of HAM-A items 1 to 6, and item 14
- Change from baseline in HAM-A somatic subscale, where the somatic subscale is the sum of HAM-A items 7 to 13

Descriptive summary statistics of baseline, HAM-A total score and change from baseline at each visit including the last assessment during treatment period will be provided by prior ALKS 5461 exposure and overall based on observed data. The HAM-A psychic subscale and somatic subscale will be summarized in a similar way. In addition, a figure of HAM-A total score (including standard error), mean change from baseline (including standard error) over time including the last assessment during treatment period will be provided by prior ALKS 5461 exposure and overall.

The individual HAM-A item score will not be summarized but will be included in the subject listing.

#### 3.6.2.3. Clinical Global Impression – Severity (CGI-S)

The CGI-S is a 7-point scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on severity of mental illness at the time of rating 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3= mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill. The rating of 0 (not assessed) will be considered as missing.

Descriptive summary statistics of baseline, CGI-S score and change from baseline at each visit including the last assessment during treatment period and follow up period will be provided by prior ALKS 5461 exposure and overall based on observed data. The number and percentage of subjects for each CGI-S category at each visit including the last assessment during treatment period and follow up period will also be summarized. In addition, figures of CGI-S score (including standard error) and mean change from baseline (including standard error)over time including the last assessment during treatment period and follow up period will be provided by prior ALKS 5461 exposure and overall based on observed data.

#### 3.7. Safety Analysis

#### 3.7.1. General Considerations

All safety endpoints will be summarized by prior ALKS 5461 exposure and overall based on observed data for the Safety Population.

#### 3.7.2. Adverse Events

Adverse events will be coded by System Organ Class and Preferred Term using the Medical Dictionary for Regulatory Activities MedDRA version 19.0. The verbatim term will be included in the AE listings. An AE will be considered as a treatment emergent adverse event (TEAE) if it starts or worsens (if present at baseline) on or after the baseline during treatment period. An AE will be considered as a PDEAE if it starts or worsens during the Post-discontinuation Safety Period which is after the last dose date plus 1 day. For the determination of TEAEs during the treatment period, AEs with the greatest severity before the baseline will be used as the benchmark for the comparison of the AEs occurring during the treatment period. For PDEAEs, the greatest severity before or on the last dose date plus 1 day will be used as the benchmark for the comparison of the AEs occurring during the Post-discontinuation Safety Period.

All AEs will be listed by subject. TEAEs / PDEAEs, deaths, serious adverse events (SAEs), AEs leading to study discontinuation will be included in the summary tables. Summary tables will be provided by prior ALKS 5461 exposure and overall for the Safety Population. For AEs leading to study discontinuation or deaths, the AEs will be summarized in the period in which the discontinuation or death occurred. Drug related TEAEs include those scored as definitely related, probably related, and possibly related by the investigator.

The following summary tables will be produced for the treatment period / Post-discontinuation Safety Period by prior ALKS 5461 exposure and overall for the Safety Population:

- Overview AE summary tables (TEAEs / PDEAEs)
- TEAEs / PDEAEs by System Organ Class and Preferred Term
- TEAEs / PDEAEs by Preferred Term in decreasing frequency
- TEAEs / PDEAEs experienced by ≥5% of subjects (in any group) by Preferred Term
- TEAEs / PDEAEs by System Organ Class, Preferred Term, and Severity
- Drug-related TEAEs by System Organ Class and Preferred Term
- SAEs (fatal and non-fatal) by System Organ Class and Preferred Term
- SAEs (fatal and non-fatal) by Preferred Term in decreasing frequency
- AEs leading to study discontinuation by System Organ Class and Preferred Term
- AEs leading to study discontinuation by Preferred Term in decreasing frequency
- TEAEs by System Organ Class, Preferred Term, and Duration of Exposure
- TEAEs by Preferred Term in decreasing frequency and Duration of Exposure
- Duration of TEAEs experienced by ≥5% of All Subjects by Preferred Term

• Incidence of TEAEs experienced by ≥5% of All Subjects by Preferred Term and Exposure Interval

A subject having the same AE (as determined by the coded MedDRA preferred term) more than once will be counted only once in the calculation of the number and percentage of subjects for that AE. Similarly, if a subject has more than one AE in a System Organ Class, the subject will be counted only once in the number of subjects with an AE for that System Organ Class. If a subject has the same AE on multiple occasions, the highest severity (severe > moderate > mild) recorded for the event will be presented in the AE by severity summary. Similarly, if a subject has the same AE on multiple occasions, the closest relationship (related > not related, where related includes definitely related, probably related, and possibly related; and not related includes probably not related and definitely not related) recorded for the event will be presented in the AE by relationship summary. If a subject has the same AE on multiple occasions, the first presentation will be used in the incidence table and the longest duration will be used in the duration table.

The number and percentage of subjects with TEAE during the ALK5461-208 study will be summarized by System Organ Class, Preferred Term, and duration of exposure since the first dose of the study drug in the ALK5461-208 study (1 day to <1 month,  $\geq$ 1 to <3 months,  $\geq$ 3 to <6 months,  $\geq$ 6 to <9 months,  $\geq$ 9 to <12 months, and  $\geq$ 12 months). For each exposure interval, the percentage will be calculated as the number of subjects with a new TEAE that started during the exposure interval, relative to the number of subjects exposed during the interval. Separate tables for prior ALKS 5461 exposure and overall will be provided.

Descriptive statistics (number of subjects, mean, SD, median, 10th percentile, 90th percentile, minimum, and maximum) of duration (days) of TEAEs experienced by ≥5% of All Subjects will be provided by Preferred Term during treatment period for the Safety Population. The duration is defined as number of days from the TEAE start date to the TEAE stop date during the ALK5461-208 study, inclusive. If a TEAE is ongoing at the end of the treatment period, the TEAE stop date is imputed by last dose date plus 1 day. For those subjects who have the same event (same PT term) that is treatment emergent on multiple occasions, we will choose the longest duration as stated above. For partial TEAE start or stop date:

- If only day is missing but month available, TEAE start date will be imputed as the first day of the month and TEAE stop date will be imputed as the last day of the month.
- If both month and day are missing, TEAE start date will be imputed as the Visit 2 date or January 1st whenever applicable, and TEAE stop date will be imputed as the last dose date or December 31st whenever applicable.

The Incidence (%) of TEAEs experienced by  $\geq 5\%$  of All Subjects by Preferred Term and Exposure Interval (1 day to <1 month,  $\geq 1$  to <3 months,  $\geq 3$  to <6 months,  $\geq 6$  to <9 months,  $\geq 9$  to <12 months, and  $\geq 12$  months) will be presented by prior ALKS 5461 exposure and overall during treatment period for the Safety Population. For those subjects who have the same event (same PT term) that is treatment emergent on multiple occasions, the first instance where that event was treatment emergent will be used, as stated above. The incidence (%) is calculated by n/m x 100%, where n is defined as the number of subjects with newly emergent or worsened adverse events during the exposure interval; m is defined as the number of subjects who had

treatment exposure during the exposure interval. The incidence (%) of TEAE over time will also be presented graphically. For each preferred term, a bar graph will be presented by prior ALKS 5461 exposure and overall. The number of n/m of three groups will be listed below the figure.

Subgroup analyses are planned for TEAEs only. Subgroups to include:

- Demographics (age [<55 years, ≥55 years], race [white, all other races], gender [female, male])
- Region (US, non-US)
- ADT class (SSRI, SNRI, and other)
- Benzodiazepines use (yes, no)
- Opioid use (yes, no)

A subject is considered as having used a Benzodiazepine (BDZ) or BDZ-like drug ("yes" subgroup) if the subject was taking any concomitant medication in the Benzodiazepine group for any duration in the treatment period of interest. A subject is considered as not having used a Benzodiazepine (BDZ) or BDZ-like drug ("no" subgroup) if the subject was not taking any concomitant medication in the Benzodiazepine group and sedating H1 antagonist group.

Similarly, a subject is considered as having used an opioid drug ("yes" subgroup) if the subject was treated with any concomitant medication in the opioid classification for any duration in the treatment period of interest. A subject is considered as not having used an opioid drug ("no" subgroup) if the subject was not treated with any concomitant medication in the opioid classification. A table of SAE by System Organ Class and Preferred Term for opioid use will be presented.

Subject listings for AEs will be included.

#### 3.7.3. Adverse Events of Special Interest

Adverse events of special interest (AESIs) will be summarized by Preferred Term and by prior ALKS 5461 exposure and overall during treatment period for the Safety Population / Post-discontinuation Safety Population for any TEAEs or PDEAEs of special interest. The following summaries will be created for AESI:

- TEAEs associated with abuse potential
- TEAEs associated with dependence
- PDEAEs associated with withdrawal
- TEAEs associated with suicidal ideation and behavior
- TEAEs associated with hypomania / mania
- TEAEs associated with central nervous system (CNS) depression and sedation
- TEAEs associated with respiratory depression
- TEAEs associated with orthostasis / hypotension
- TEAEs associated with hypersensitivity

- TEAEs associated with slowing of ventricular repolarization
- TEAEs associated with hepatic effects
- TEAEs associated with sexual dysfunction

TEAEs associated with abuse potential will be presented by Adhoc System Organ Class and Preferred Term, where Adhoc System Organ Class is manually classified by Alkermes medical director as 3 categories: abuse behavior, euphoria related, and non-specific.

TEAEs associated with dependence will be presented for subjects with any exposure, ≥4 weeks exposure, and <4 weeks exposure, respectively.

PDEAEs associated with withdrawal will be presented for subjects with any exposure, ≥4 weeks exposure, and <4 weeks exposure, respectively. AESIs associated with withdrawal are PDEAEs that occur from >2 to 16 days post last dose as this is the period during which physiological opioid withdrawal presents by considering half-lives of both BUP and SAM.

Supportive AE listings will be provided for each special interest group. Narratives will be provided for clinically meaningful events within each AESI group.

#### 3.7.4. Clinical Laboratory Parameters

Laboratory parameters will be presented in conventional units. Only scheduled laboratory assessments will be included in the summaries of mean and change from baseline descriptive analyses. Laboratory assessments from both scheduled and unscheduled visits will be included in outlier analyses. Outlier analyses will not include post-discontinuation assessments. All laboratory data will be included in the listings. Parameter order for summary tables and listings will be by system (renal, hepatic, etc.).

#### 3.7.4.1. Descriptive Analysis of Laboratory Parameters

Numerical laboratory results (baseline and change from baseline) for chemistry and hematology parameters and urinalysis (pH and Specific Gravity) for each visit during the entire study (including last assessment during treatment period and visits in Post-discontinuation Safety Period) will be summarized (number of subjects, mean, SD, median, minimum, and maximum) by prior ALKS 5461 exposure and overall for the Safety Population.

In addition, baseline and post-baseline observed values (lowest, highest, last assessment during treatment period), and change from baseline to lowest, highest and last assessment values during the treatment period for chemistry and hematology parameters, urinalysis (pH and Specific Gravity), will be summarized by prior ALKS 5461 exposure and overall for the Safety Population.

The following graphical displays for laboratory parameters (chemistry, hematology, and urinalysis) will be presented during the entire study (including last assessment during treatment period and Post-discontinuation Safety Period) by prior ALKS 5461 exposure and overall for the Safety Population:

- Line graphs for mean change from baseline along with the corresponding standard error (SE; including Post-discontinuation Safety Period)
- Box-and-Whisker figures for baseline and post-baseline observed values (lowest, highest, last assessment during treatment period)
- Box-and-Whisker figures for change from baseline to the lowest post-baseline value, the highest post-baseline value, and the last scheduled post-baseline value during treatment period
- Scatter plots for baseline and post-baseline observed values (lowest, highest, last assessment during treatment period)

#### 3.7.4.2. Outlier Analyses of Laboratory Parameters

The number and percentage of subjects with values considered potentially clinically significant (PCS) occurring at any post-baseline visit during treatment period for selected parameters will be summarized. For PCS, the summary will be provided by prior ALKS 5461 exposure and overall for the Safety Population. These analyses do not include Post-discontinuation Safety Period.

Clinical laboratory test values, scheduled or unscheduled, will be considered PCS if they meet the PCS criteria listed in Table 4. The percentage will be calculated relative to the number of subjects with available non-PCS baseline values with respect to the specific criterion and at least 1 post-baseline assessment. The numerator is the total number of subjects with a non-PCS baseline value with respect to the specific criterion and at least 1 post-baseline PCS value. A supportive listing will present all values for a parameter for subjects with at least 1 PCS value for that parameter.

Shift tables for shift from within normal reference limits / high to low and shift from within normal reference limits / low to high during treatment period will be provided for chemistry, hematology, and urinalysis parameters with conventional reference limits (limits provided by the performing laboratories) by prior ALKS 5461 exposure and overall for the Safety Population. For parameters which have gender and / or age specific limits, the categories will be based on the specific limits. High is defined as values greater than the upper limit of the reference range (ULRR). Low is defined as values less than the lower limit of the reference range (LLRR). Normal reference limits is defined as values within normal range. The analysis population consists of subjects in the Safety Population with a baseline value outside the specific shift direction. All laboratory values collected during the treatment period will be considered in this analysis.

The percentages will be calculated for the shift summary as follows:

- For the shifts from within normal reference limits / high to low: the numerator is defined as the number of subjects with a post-baseline result below the LLRR, and the denominator is defined as the number of subjects with a baseline value within the limits or above the ULRR.
- For the shifts from within normal reference limits / low to high: the numerator is defined as the number of subjects with a post-baseline results above the ULRR, and the denominator is defined as the number of subjects with a baseline value within the limits or below the LLRR.

Pregnancy and drug screening data will be listed. For urinalysis, rate of abnormalities at any post-baseline visit during treatment period will be summarized.

 Table 4:
 Potentially Clinically Significant Abnormal Laboratory Values

| Category | Parameter | Criteria |
|---|---|---|
| Hematology | Eosinophils | $>1.0x10^3/\mu L$ |
| | Hematocrit | ≤32% and 3 point decrease from baseline (Female)<br>≤37% and 3 point decrease from baseline (Male) |
| | Hemoglobin | ≤9.5 g/dL (Female)<br>≤11.5 g/dL (Male) |
| | Leukocytes | $\leq 2.8 \times 10^{3} / \mu L$<br>$\geq 16 \times 10^{3} / \mu L$ |
| | Neutrophils, Absolute | $<1.5x10^{3}/\mu L$ |
| | Platelets | $<75.1 \times 10^{3} / \mu L$<br>$\geq 700 \times 10^{3} / \mu L$ |
| Chemistry | Alanine Aminotransferase | ≥3xULRR |
| | Albumin | <2.5 g/dL |
| | Alkaline Phosphatase | ≥3xULRR |
| | Aspartate Aminotransferase | ≥3xULRR |
| | Bicarbonate | <15 mmol/L<br>>31 mmol/L |
| | Blood Urea Nitrogen (BUN) | >30 mg/dL |
| | Calcium | <8.2 mg/dL<br>>12 mg/dL |
| | Chloride | ≤90 mmol/L<br>≥118 mmol/L |
| | Creatine Phosphokinase | >3xULRR |
| | Creatinine | ≥2 mg/dL |

Table 4: Potentially Clinically Significant Abnormal Laboratory Values (Continued)

| Category | Parameter | Criteria |
|---|---|---|
| | Gamma Glutamyltransferase | ≥3xULRR |
| | Glucose | <50 mg/dL |
| | | >200 mg/dL |
| | HDL Cholesterol | ≤30 mg/dL |
| | Lactate Dehydrogenase | >3xULRR |
| | LDL Cholesterol | ≥160 mg/dL |
| | Phosphate | <2 mg/dL<br>>5 mg/dL |
| | Potassium | <3 mmol/L<br>>5.5 mmol/L |
| | Prolactin | >1xULRR |
| | Sodium | <130 mmol/L<br>>150 mmol/L |
| | Total Bilirubin | ≥2 mg/dL |
| | Total Cholesterol | >300 mg/dL |
| | Triglycerides | ≥120 mg/dL (Female)<br>≥160 mg/dL (Male) |
| | Uric Acid | >9 mg/dL<br>>8 mg/dL (Female)<br>>10 mg/dL (Male) |
| Urinalysis | Glucose<br>Protein | at least 2+ |

Abbreviations: BUN=blood urea nitrogen; HDL=high density lipoproteins; LDL=low density lipoprotein; ULRR=upper limit of referene range

#### 3.7.4.3. Hepatic Effects

Analyses on hepatic analytes will be performed on some laboratory measures to assess potential hepatic effects and will include alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin (TBILI). Hepatic effects will be explored using drug induced liver injury (DILI) criteria from the FDA guidance as well as Hy's Law criteria and through individual frequencies of abnormalities compared to reference limits. Summaries will be presented by prior ALKS 5461 exposure and overall for the Safety Population. DILI and Hy's Law criteria are defined relative to the ULRR as follows:

- $((ALT \text{ or } AST) \ge 3xULRR) \& (TBILI \ge 1.5xULRR)$
- $((ALT \text{ or } AST) \ge 3xULRR) \& (TBILI \ge 1.5xULRR) \& (ALP < 2xULRR)$
- $((ALT \text{ or } AST) \ge 3xULRR) \& (TBILI \ge 2xULRR)$
- $((ALT \text{ or } AST) \ge 3xULRR) \& (TBILI \ge 2xULRR) \& (ALP < 2xULRR)$

To complement the DILI and Hy's Law analyses described above, an "evaluation of drug-induced serious hepatotoxicity" (eDISH) plot will present maximum TBILI versus maximum ALT / AST by study group during treatment period for the Safety Population. Individual subject values for the maximum ALT / AST value expressed as the multiple of the ULRR versus the maximum TBILI value also expressed as the multiple of the ULRR will be presented. Reference lines will indicate values that fall within the range of DILI or Hy's Law criteria.

The listing of subjects meeting the DILI or Hy's Law citeria with all values of relevant laboratory parameters will be provided.

The number and percentage of subjects with certain baseline values for ALT, AST, TBILI and who have any post-baseline values meeting the shift criteria specified in Table 5, Table 6 and Table 7 during treatment period will be summarized, respectively. The numerator is the number of subjects with baseline meeting the specific baseline criterion and at least 1 post-baseline assessment. The denominator is the number of subjects with baseline meeting the specific baseline criterion and at least 1 post-baseline ALT / AST / TBILI elevation value.

Table 5: Shift Criteria and Denominator for Alanine Aminotransferase (ALT)

| | Denominator | | |
|---|---|---|---|
| ALT Elevations During Treatment Period | All Subjects | Subjects with Baseline<br>Values ≤1xULRR | Subjects with Baseline<br>Values >1xULRR |
| ≥3xULRR | Baseline <3xULRR | | Baseline >1xULRR |
| ≥5xULRR | Baseline <5xULRR | Dagalina /1vIII DD | |
| ≥10xULRR | Baseline <10xULRR | Baseline ≤1xULRR | |
| ≥20xULRR | Baseline <20xULRR | | |

Abbreviations: ULRR=upper limit of reference range

Table 6: Shift Criteria and Denominator for Aspartate Aminotransferase (AST)

| | Denominator | | |
|---|---|---|---|
| AST Elevations During Treatment Period | All Subjects | Subjects with Baseline<br>Values ≤1xULRR | Subjects with Baseline<br>Values >1xULRR |
| ≥3xULRR | Baseline <3xULRR | | Baseline >1xULRR |
| ≥5xULRR | Baseline <5xULRR | Dagalina / LyLIL DD | |
| ≥10xULRR | Baseline <10xULRR | Baseline ≤1xULRR | |
| ≥20xULRR | Baseline <20xULRR | | |

Abbreviations: ULRR=upper limit of reference range

Table 7: Shift Criteria and Denominator for Total Bilirubin (TBILI)

| Total Bilirubin Elevations During<br>Treatment Period | Denominator |
|---|---|
| ≥2xULRR | All Subjects with Baseline <2xULRR |
| ≥2xULRR | Baseline ≤1xULRR |
| ≥2xBaseline | Baseline >1xULRR |

Abbreviations: ULRR=upper limit of reference range

#### 3.7.5. Vital Signs

Vital signs (supine systolic and supine diastolic blood pressure, heart rate, respiratory rate, temperature, weight, and BMI) will be summarized for baseline and change from baseline (BMI baseline only) by prior ALKS 5461 exposure and overall for the Safety Population, and will include post-discontinuation assessments.

In addition, baseline and post-baseline observed values (lowest, highest, last assessment during treatment period), and change from baseline to lowest, highest and last assessment values during treatment period for vital sign parameters will be summarized by prior ALKS 5461 exposure and overall for the Safety Population, and will not include post-discontinuation assessments.

The following graphical displays for vital sign parameters will be presented by prior ALKS 5461 exposure and overall for the Safety Population:

- Line graphs for mean change from baseline along with the corresponding SE (including Post-discontinuation Safety Period)
- Box-and-Whisker figures for baseline and post-baseline observed values (lowest, highest, and last assessment during treatment period)
- Box-and-Whisker figures for change from baseline to the lowest post-baseline value, the highest post-baseline value, and the last scheduled post-baseline value during treatment period
- Scatter plots for baseline and post-baseline observed values (lowest, highest, and last assessment during treatment period)

Vital signs will also be evaluated using PCS criteria as indicated in Table 8 and summarized by prior ALKS 5461 exposure and overall for the Safety Population. Post-discontinuation assessments will not be included in this analysis.

 Table 8:
 Potentially Clinically Significant Abnormal Vital Sign Values

| Parameter | PCS Criteria |
|---------------------------------|-----------------------------------------|
| Temperature | Hyperthermia: ≥38.1°C |
| | Hypothermia: ≤35.0°C |
| Supine Systolic Blood Pressure | Low: ≤90 mm Hg and decrease ≥20 mm Hg |
| | High: ≥140 mm Hg and increase ≥20 mm Hg |
| Supine Diastolic Blood Pressure | Low: ≤50 mm Hg and decrease ≥10 mm Hg |
| | High: ≥90 mm Hg and increase ≥10 mm Hg |
| Heart Rate | Low: ≤50 bpm and decrease ≥15 bpm |
| | High: ≥100 bpm and increase ≥15 bpm |
| Respiratory Rate | Low: <12 breaths per minute |
| | High: >25 breaths per minute |
| Body Weight | Decrease from baseline ≥7% |
| | Increase from baseline ≥7% |

A supportive listing will present for subjects and parameter for cases where at least 1 value was potentially significant.

#### 3.7.6. Electrocardiograms

Electrocardiogram (ECG) parameters (heart rate, RR interval, PR interval, QRS interval, QT interval, and QTcF [QT interval corrected using Fridericia's method]) will be summarized (baseline and change from baseline) for each visit during the entire study, including last assessment during treatment period and post-discontinuation assessments.

In addition, baseline and post-baseline observed values (lowest, highest, last assessment during treatment period), and change from baseline to lowest, highest and last assessment values during treatment period for ECG parameters will be summarized by prior ALKS 5461 exposure and overall for the Safety Population. These analyses will not include post-discontinuation values.

The following graphical displays for ECG will be presented by prior ALKS 5461 exposure and overall for the Safety Population:

- Line graphs for mean change from baseline along with the corresponding SE (including Post-discontinuation Safety Period)
- Box-and-Whisker figures for baseline and post-baseline observed values (lowest, highest, last assessment during treatment period)
- Box-and-Whisker figures for change from baseline to the lowest post-baseline value, the highest post-baseline value, and the last scheduled post-baseline value during treatment period
- Scatter plots for baseline and post-baseline observed values (lowest, highest, last assessment during treatment period)

ECG will be evaluated using PCS criteria as indicated in Table 9 by prior ALKS 5461 exposure and overall for the Safety Population. These analyses will not include post-discontinuation assessments.

 Table 9:
 Potentially Clinically Significant Abnormal ECG Values

| ECG Parameter | PCS Criteria |
|---------------|---------------------------------------------------------|
| PR Interval | High: ≥220 msec |
| QRS Interval | High: ≥120 msec |
| QTcF | Low: <330 msec<br>High: >450 msec; >480 msec; >500 msec |
| | Only cumulative incidence above the indicated limits |
| QTcF | Change from baseline increase/decrease >30 msec |
| | Change from baseline increase/decrease >60 msec |
| Heart Rate | Low: ≤50 bpm and decrease ≥15 bpm |
| | High: ≥100 bpm and increase ≥15 bpm |

A supportive listing will present all values for a parameter for subjects with at least 1 PCS value for that parameter.

#### 3.7.7. Columbia Suicide Severity Rating Scale (C-SSRS)

Columbia Suicide Severity Rating Scale items of suicidal behavior and suicidal ideation will be summarized at baseline and post-baseline by prior ALKS 5461 exposure and overall for the Safety Population. The proportion of subjects who meet the criterion for each of these categories will be summarized as described in Table 10. Each item will be presented separately within each category (suicidal behavior, suicidal ideation, self-injurious behavior without suicidal intent). Any suicide attempt (aborted, interrupted, and actual) will also be summarized as a category. Data will be presented for baseline, any post-baseline (i.e. on treatment), and any post-discontinuation values.

Any behaviors experienced will be listed with a brief narrative. Any completed suicides will be presented with full narrative.

**Table 10:** C-SSRS Summary Categories for Analysis

| Category | C-SSRS item response is "YES" |
|---|---|
| Suicidal ideation | 1) Wish to be dead |
| | 2) Non-specific active suicidal thoughts |
| | 3) Active suicidal ideation with any methods (not plan) without intent to act |
| | 4) Active suicidal ideation with some intent to act, without specific plan |
| | 5) Active suicidal ideation with specific plan and intent |
| Suicidal behavior | 6) Preparatory acts or behavior |
| | 7) Aborted attempt |
| | 8) Interrupted attempt |
| | 9) Actual attempt |
| | 10) Completed suicide |
| Suicidal behavior or ideation | Including 10 items above |
| Self-injurious behavior without suicidal intent | Purely for other reasons / without any intention of killing yourself |

Summary of treatment emergent suicide-related events based on the C-SSRS during treatment period will be presented by prior ALKS 5461 exposure and overall for the Safety Population. The degree and type of treatment emergent suicide-related events will be summarized in a table as defined in Table 11. Post-discontinuation assessments will not be included in this analysis.

This analysis population consists of safety population with non-missing baseline and at least 1 post-baseline assessment during treatment period. The percentage will be calculated for the treatment emergent suicide-related event summary. The numerator is defined as the number of subjects with a non-missing baseline and a post-baseline C-SSRS assessment meeting the treatment emergent suicide-related numerator criteria defined in Table 11, and the denominator is defined as the number of subjects with a non-missing baseline and at least 1 post-baseline C-SSRS assessment meeting the treatment emergent suicide-related denominator criteria defined in Table 11 during treatment period.

**Table 11:** Treatment Emergent Suicide-related Events for Analysis

| Treatment Emergent Suicide-<br>related Events | Denominator Criteria | Numerator Criteria |
|---|---|---|
| Increase in Suicidal Ideation from Baseline | Baseline suicidal ideation ("No" to all ideation items 1- 5, or "Yes" to any ideation item ≤4 and "No" to item 5) | Baseline suicidal ideation ("No" to all ideation items 1-5, or "Yes" to any ideation item ≤4 and "No" to item 5) |
| | | Post-baseline (increase in suicidal ideation severity from baseline at any post-baseline visit) |
| Emergence of Serious Suicidal Ideation | Baseline suicidal ideation<br>("No" to all ideation items 1-<br>5, or "Yes" to any ideation<br>item≤3 and "No" to items 4<br>and 5) | Baseline suicidal ideation ("No" to all ideation items 1-5, or "Yes" to any ideation item ≤3 and "No" to items 4 and 5) Post-baseline ("Yes" to ideation item 4 or 5 at any post-baseline visit) |
| Emergence of Serious Suicidal<br>Ideation in Subjects with no<br>Suicidal Ideation at Baseline | Baseline ideation ("No" to all ideation items 1-5) | Baseline ideation ("No" to all ideation items 1-5) Post-baseline ("Yes" to ideation item 4 or 5 at any post-baseline visit) |
| Decrease in Suicidal Ideation from Baseline | Baseline ideation ("Yes" to any ideation items 1-5) | Baseline ideation ("Yes" to any ideation items 1-5) Post-baseline (decrease in suicidal ideation severity at any post-baseline visit compared to severity at baseline) |
| Emergence of Suicidal Behavior in<br>Subjects with no Suicidal Behavior<br>at Baseline | Baseline behavior ("No" to all behavior items 6-10) | Baseline behavior ("No" to all behavior items 6-10) Post-baseline behavior ("Yes" to any behavior items 6-10 at any post-baseline visit) |

#### 3.7.8. Clinical Opiate Withdrawal Scale (COWS) Scores

COWS will be administered only at EOT and post-discontinuation visits, so COWS will be analyzed for Post-discontinuation Safety Population. For Post-discontinuation Safety Population, baseline COWS is defined as EOT COWS assessment. Adequate COWS baseline is defined as EOT COWS assessment being performed within ( $\leq$ ) 2 days of last dose of study drug.

Subjects will be included in the COWS analysis if they have an adequate EOT COWS and at least 1 post-EOT COWS in the post-discontinuation safety period. COWS will be summarized by:

- Analysis of all post-EOT COWS assessments
- Analysis of post-EOT COWS assessments that occurred from >2 to 16 days post last dose of study drug

Subjects with inadequate EOT COWS, i.e. EOT COWS assessment was performed more than (>) 2 days of last dose, will be included in a supportive listing.

Although opioid withdrawal might not be expected in individuals with less than 4 weeks of drug exposure, COWS will be presented in all subjects with adequate EOT COWS, and then COWS will be subset by duration of study drug exposure. Three COWS analyses will be presented for the subjects with adequate EOT COWS by the 3 exposure subgroups (any exposure, ≥4 weeks exposure, <4 weeks exposure):

- Total COWS scores (baseline and change from baseline, and days between last dose and assessment date) will be summarized by visit (baseline, post-discontinuation visits)
- Subject count and incidence will be provided by visit for each of the COWS total score categories indicated below:

No withdrawal: total score 0-4

Mild withdrawal: total score 5-12

Moderate withdrawal: total score 13-24

Moderately severe withdrawal: total score 25-36

- Severe withdrawal: total score >36

COWS category shift summary from baseline to post-baseline: the numerator is the
number of subjects in each post-discontinuation COWS category with non-missing
baseline COWS. If there are more than one post-discontinuation COWS, i.e. a subject
with an unscheduled visit, the highest value will be used. The denominator is the
number of subjects in each baseline COWS category.

Data listing of COWS scores at each visit will be provided. Narratives will be provided for any clinically meaningful COWS shifts.

#### 4. INTERIM ANALYSES

No interim analysis is planned.

# 5. CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL

N/A.

# 6. DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA

Dataset specifications will be provided in a separate document.

# **6.1.** Analysis Visit Windows

Every attempt must be made to provide complete data. In cases where complete data cannot be collected, the principles to assign the analysis visits for inclusion in summary tables described in this section will be followed for data handling and analyses.

Early termination visits for efficacy measurements will be mapped to the next scheduled visit. For example, a subject who terminates shortly after Day 29 (e.g., has assessments at baseline through Day 29, and Day 365 or early termination) would have assessments at early termination mapped to the next scheduled visit for each assessment. In this example, the MADRS and CGI-S from the early termination visit would be mapped to Day 43; and the HAM-A results would be mapped to Day 57. For other visits other than early termination / Day 365, the visit number indicated on the CRF (i.e., CRF visit) will be used as the analysis visit.

Early termination visits for safety measurements will not be mapped to any scheduled post-baseline visit, but will be used as the last assessment during treatment period.

Measurements collected from unscheduled visits will not be included in the by-visit summary tables or mean change analyses but will be included in the analysis of outlier and PCS values and in the subject listings.

# 6.2. Efficacy Data Handling

MADRS-10 is the sum of the 10 items from the MADRS. HAM-A total score is the sum of 14 items from the HAM-A. If only one of the items of the MADRS, or HAM-A for a given visit is missing, then the total score will be calculated using (sum of non-missing items) × (total number of items) / (number of non-missing items). If more than one of the items are missing, the total score will be set to missing. The MADRS-6 and HAM-A subscale scores will be set to missing if any item is missing.

#### 6.3. Handling of Partial Dates of Prior and Concomitant Medications

Partial start dates of prior and concomitant medications will be assumed to be the earliest possible date consistent with the partial date. Partial stop dates of prior and concomitant medications will be assumed to be the latest possible date consistent with the partial date. In the case of completely missing stop date, medication will be assumed to be ongoing.

#### 7. GENERAL STATISTICAL METHODOLOGY

#### 7.1. Statistical Conventions

In general, summary statistics (n, mean, standard deviation [SD], median, minimum and maximum for continuous variables, and number and percentage of subjects in each category for categorical variables) will be provided by study group. All summary tables will be based on observed data, and missing values will not be imputed unless otherwise indicated. Measurements collected from unscheduled visits or repeated assessments will not be included in the by-visit summary or mean change tables or figures, but will be included in the analyses for the outlier / PCS post-baseline values, and subject listings. Source data for the summary tables and statistical analyses will be presented as subject data listings.

# 7.2. Reporting Precision

Summary statistics will be presented to the degree of precision in Table 12, unless otherwise specified.

**Table 12:** Degree of Precision

| Statistics | Degree of Precision |
|---|---|
| Mean, Median, Quartiles, Confidence | One more than the raw data, up to 3 decimal places. |
| limit boundaries | |
| Standard deviation, Standard error | One more than the mean, up to 3 decimal places. |
| Minimum, Maximum | The same as the raw data. |
| p-value | Rounded to 3 decimal places and therefore presented |
| | as 0.xxx; p-values smaller than 0.001 as '<0.001'; p- |
| | values greater than 0.999 as '>0.999'. |
| Percentage | One decimal place. A percentage of 100% will be |
| | reported as 100%. Percentages of zero will be |
| | reported as 0. |

Fractional numeric values will be presented with a zero to the left of the decimal point (for example, 0.12–0.30).

For weight, height, and BMI, one decimal place will be used for summary statistics.

## 8. PROGRAMMING SPECIFICATIONS

Programming specifications will be provided in a separate document.

# 9. MOCK TABLES, LISTINGS AND FIGURES (TLFS)

Mock-up tables, listings, and figures will be provided in a separate document.

# 10. REFERENCES

1. Alkermes ALK5461-208 Study Protocol Amendment 3 (dated 03 March 2016).

# APPENDIX 1. AESI – ABUSE POTENTIAL

| Preferred Term | Adhoc SOC |
|-----------------------------------------------|-------------------|
| Accidental overdose | AP_abuse behavior |
| Drug abuser | AP_abuse behavior |
| Drug diversion | AP_abuse behavior |
| Drug level above therapeutic | AP_abuse behavior |
| Drug level increased | AP_abuse behavior |
| Drug screen | AP_abuse behavior |
| Drug screen positive | AP_abuse behavior |
| Intentional overdose | AP_abuse behavior |
| Intentional product misuse | AP_abuse behavior |
| Intentional product use issue | AP_abuse behavior |
| Maternal use of illicit drugs | AP_abuse behavior |
| Needle track marks | AP_abuse behavior |
| Neonatal complications of substance abuse | AP_abuse behavior |
| Overdose | AP_abuse behavior |
| Prescription drug used without a prescription | AP_abuse behavior |
| Prescription form tampering | AP_abuse behavior |
| Product tampering | AP_abuse behavior |
| Substance abuse | AP_abuse behavior |
| Substance abuser | AP_abuse behavior |
| Substance use | AP_abuse behavior |
| Substance-induced mood disorder | AP_abuse behavior |
| Substance-induced psychotic disorder | AP_abuse behavior |
| Toxicity to various agents | AP_abuse behavior |
| Acute psychosis | AP_non-specific |
| Aggression | AP_non-specific |
| Cognitive disorder | AP_non-specific |
| Confusional state | AP_non-specific |
| Delirium | AP_non-specific |
| Delusional disorder, unspecified type | AP_non-specific |
| Depersonalisation/derealisation disorder | AP_non-specific |
| Disorientation | AP_non-specific |
| Dissociation | AP_non-specific |
| Disturbance in attention | AP_non-specific |
| Disturbance in social behaviour | AP_non-specific |
| Dizziness | AP_non-specific |
| Dopamine dysregulation syndrome | AP_non-specific |
| Emotional disorder | AP_non-specific |
| Flight of ideas | AP_non-specific |
| Medication overuse headache | AP_non-specific |
| Preferred Term | Adhoc SOC |
|-----------------------------|---------------------|
| Mental impairment | AP_non-specific |
| Mood altered | AP_non-specific |
| Mood swings | AP_non-specific |
| Narcotic bowel syndrome | AP_non-specific |
| Paranoia | AP_non-specific |
| Psychotic behaviour | AP_non-specific |
| Psychotic disorder | AP_non-specific |
| Sedation | AP_non-specific |
| Somnolence | AP_non-specific |
| Stupor | AP_non-specific |
| Euphoric mood | AP-euphoria related |
| Feeling abnormal | AP-euphoria related |
| Feeling drunk | AP-euphoria related |
| Feeling of relaxation | AP-euphoria related |
| Hallucination | AP-euphoria related |
| Hallucination, auditory | AP-euphoria related |
| Hallucination, gustatory | AP-euphoria related |
| Hallucination, mixed | AP-euphoria related |
| Hallucination, olfactory | AP-euphoria related |
| Hallucination, synaesthetic | AP-euphoria related |
| Hallucination, tactile | AP-euphoria related |
| Hallucination, visual | AP-euphoria related |
| Inappropriate affect | AP-euphoria related |
| Thinking abnormal | AP-euphoria related |

# APPENDIX 2. AESI – DEPENDENCE

| Preferred Term |
|-----------------------------|
| Dependence |
| Drug dependence |
| Drug dependence, antepartum |
| Drug dependence, postpartum |
| Drug tolerance |
| Drug tolerance decreased |
| Drug tolerance increased |
| Substance dependence |

# APPENDIX 3. AESI – WITHDRAWAL

| Drug detoxification Reversal of opiate activity Drug rehabilitation Drug withdrawal convulsions Drug withdrawal headache Drug withdrawal maintenance therapy Drug withdrawal syndrome Drug withdrawal syndrome neonatal |
|---|
| Drug rehabilitation Drug withdrawal convulsions Drug withdrawal headache Drug withdrawal maintenance therapy Drug withdrawal syndrome |
| Drug withdrawal convulsions Drug withdrawal headache Drug withdrawal maintenance therapy Drug withdrawal syndrome |
| Drug withdrawal headache Drug withdrawal maintenance therapy Drug withdrawal syndrome |
| Drug withdrawal maintenance therapy Drug withdrawal syndrome |
| Drug withdrawal syndrome |
| Drug withdrawal syndrome neonatal |
| Rebound effect |
| Steroid withdrawal syndrome |
| Withdrawal arrhythmia |
| Withdrawal syndrome |
| Anhedonia |
| Depressed mood |
| Depression |
| Dysphoria |
| Feeling of despair |
| Morose |
| Negative thoughts |
| Persistent depressive disorder |
| Dyssomnia |
| Headache |
| Insomnia |
| Obsessive thoughts |
| Poor quality sleep |
| Syncope |
| Terminal insomnia |
| Agitation |
| Irritability |
| Anxiety |
| Chills |
| Hyperhidrosis |
| Nausea |
| Nervousness |
| Pain |
| Tremor |
| Vomiting |
| Abdominal pain |
| Arthralgia |

| Preferred Term |
|----------------|
| Diarrhoea |
| Mydriasis |
| Piloerection |
| Restlessness |
| Rhinorrhoea |
| Tachycardia |
| Yawning |

### APPENDIX 4. AESI – SUICIDAL IDEATION AND BEHAVIOR

| Preferred Term |
|-------------------------------------------------|
| Depression suicidal |
| Suicidal ideation |
| Suicide threat |
| Suicidal behavior |
| Suicide attempt |
| Intentional overdose |
| Multiple drug overdose |
| Multiple drug overdose intentional |
| Overdose |
| Poisoning deliberate |
| Completed suicide |
| Intentional self-injury |
| Self injurious behavior |
| Self mutilation |
| Self-injurious ideation |
| Columbia suicide severity rating scale abnormal |

### APPENDIX 5. AESI – HYPOMANIA/MANIA

| Affective ambivalence Affect lability Agitation Aggression |
|------------------------------------------------------------|
| Agitation |
| Aggression |
| Anger |
| Bipolar disorder |
| Bipolar I disorder |
| Bipolar II disorder |
| Cyclothymic disorder |
| Delusion |
| Energy increased |
| Euphoric mood |
| Flight of ideas |
| Frustration tolerance decreased |
| Grandiosity |
| Hallucination |
| Hostility |
| Hypomania |
| Inappropriate affect |
| Irritability |
| Mania |
| Mood swings |
| Sexually inappropriate behavior |

### APPENDIX 6. AESI – CNS DEPRESSION AND SEDATION

| Preferred Term |
|-------------------------------------------------------------------|
| Apathy |
| Asthenia |
| Bradyphrenia |
| Decreased activity |
| Decreased interest |
| Depressed level of consciousness |
| Fatigue |
| Hypersomnia |
| Hypersomnia related to another mental condition |
| Hypokinesia neonatal |
| Hyporesponsive to stimuli |
| Hypotonic-hyporesponsive episode |
| Lethargy |
| Listless |
| Loss of consciousness |
| Neonatal oversedation |
| Prostration |
| Psychomotor retardation |
| Sedation |
| Sense of oppression |
| Sleep disorder due to general medical condition, hypersomnia type |
| Sluggishness |
| Somnolence |
| Somnolence neonatal |
| Sopor |
| Unresponsive to stimuli |

### APPENDIX 7. AESI – RESPIRATORY DEPRESSION

| Preferred Term |
|-----------------------------------|
| Acute respiratory failure |
| Apnoea |
| Apnoeic attack |
| Bradypnoea |
| Breath holding |
| Breath sounds abnormal |
| Breath sounds absent |
| Central-alveolar hypoventilation |
| Hypopnoea |
| Hypoventilation |
| Hypoventilation neonatal |
| Infantile apnoea |
| Lung hypoinflation |
| Neonatal respiratory arrest |
| Neonatal respiratory depression |
| Neonatal respiratory failure |
| Postoperative respiratory failure |
| Respiratory arrest |
| Respiratory depression |
| Respiratory depth decreased |
| Respiratory failure |
| Respiratory paralysis |
| Respiratory rate decreased |

### APPENDIX 8. AESI – ORTHOSTASIS HYPOTENSION

| Autonomic nervous system imbalance Blood pressure abnormal Blood pressure ambulatory decreased Blood pressure decreased Blood pressure diastolic abnormal Blood pressure diastolic abnormal Blood pressure diastolic abnormal Blood pressure fluctuation Blood pressure fluctuation Blood pressure remeasurable Blood pressure orthostatic Blood pressure orthostatic Blood pressure orthostatic Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock Symptom Syncope | Preferred Term |
|---|---|
| Blood pressure ambulatory abnormal Blood pressure ambulatory decreased Blood pressure decreased Blood pressure diastolic abnormal Blood pressure diastolic decreased Blood pressure fluctuation Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Preseyncope Presedural hypotension Shock Shock symptom | Autonomic nervous system imbalance |
| Blood pressure ambulatory decreased Blood pressure decreased Blood pressure diastolic abnormal Blood pressure diastolic decreased Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic pressure systolic abnormal Blood pressure systolic abn | Blood pressure abnormal |
| Blood pressure diastolic abnormal Blood pressure diastolic decreased Blood pressure idiastolic decreased Blood pressure inmeasurable Blood pressure orthostatic Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure decreased Mean arterial pressure decreased Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure ambulatory abnormal |
| Blood pressure diastolic abnormal Blood pressure diastolic decreased Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic decreased Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Creptional circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure ambulatory decreased |
| Blood pressure diastolic decreased Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness postural Hypoperfusion Hypotension Hypotension Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Presyncope Procedural hypotension Shock Shock symptom | Blood pressure decreased |
| Blood pressure fluctuation Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness postural Hypoperfusion Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure diastolic abnormal |
| Blood pressure immeasurable Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure diastolic decreased |
| Blood pressure orthostatic Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Procedural hypotension Shock Shock Shock Symptom | Blood pressure fluctuation |
| Blood pressure orthostatic decreased Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure immeasurable |
| Blood pressure systolic abnormal Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock Shock symptom | Blood pressure orthostatic |
| Blood pressure systolic decreased Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure orthostatic decreased |
| Circulatory collapse Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock Shock symptom | Blood pressure systolic abnormal |
| Circulatory failure neonatal Diastolic hypotension Dizziness exertional Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Blood pressure systolic decreased |
| Diastolic hypotension Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Circulatory collapse |
| Dizziness exertional Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Circulatory failure neonatal |
| Dizziness Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Diastolic hypotension |
| Dizziness postural Hypoperfusion Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Dizziness exertional |
| Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Precedural hypotension Shock Shock symptom | Dizziness |
| Hypotension Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Dizziness postural |
| Labile blood pressure Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Hypoperfusion |
| Mean arterial pressure decreased Neonatal hypotension Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | |
| Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Labile blood pressure |
| Neurogenic shock Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Mean arterial pressure decreased |
| Orthostatic heart rate response increased Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Neonatal hypotension |
| Orthostatic hypotension Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Neurogenic shock |
| Orthostatic intolerance Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Orthostatic heart rate response increased |
| Peripheral circulatory failure Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Orthostatic hypotension |
| Postural orthostatic tachycardia syndrome Presyncope Procedural hypotension Shock Shock symptom | Orthostatic intolerance |
| Presyncope Procedural hypotension Shock Shock symptom | Peripheral circulatory failure |
| Procedural hypotension Shock Shock symptom | Postural orthostatic tachycardia syndrome |
| Shock symptom | · · |
| Shock symptom | Procedural hypotension |
| · | Shock |
| Syncope | Shock symptom |
| | Syncope |

### APPENDIX 9. AESI – HYPERSENSITIVITY

| Acute generalised exanthematous pustulosis Acute haemorrhagic oedema of infancy Administration site dermatitis Administration site eczema Administration site hypersensitivity Administration site rash Administration site urticaria Administration site urticaria Administration site urticaria Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic coystitis Allergic cystitis Allergic gastroenteritis Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic hepatitis Allergic hepatitis Allergic oedema Allergic otitis externa Allergic otitis media Allergic otitis media Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis |
|---|
| Administration site dermatitis Administration site ezema Administration site hypersensitivity Administration site rash Administration site recall reaction Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic coystitis Allergic gestroenteritis Allergic gastroenteritis Allergic granulomatous angiitis Allergic granulomatous angiitis Allergic from yocarditis Allergic from yocarditis Allergic odema Allergic otitis externa Allergic respiratory disease Allergic respiratory symptom Allergic respiratory symptom Allergic respiratory necction |
| Administration site eczema Administration site hypersensitivity Administration site rash Administration site recall reaction Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic coystitis Allergic essinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic keratitis Allergic hepatitis Allergic hepatitis Allergic wyocarditis Allergic otitis externa Allergic otitis externa Allergic otitis externa Allergic otitis media Allergic prayngitis Allergic prayngitis Allergic respiratory disease Allergic respiratory symptom Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic respiratory reaction |
| Administration site hypersensitivity Administration site rash Administration site recall reaction Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic cosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic keratitis Allergic hepatitis Allergic wyocarditis Allergic myocarditis Allergic oedema Allergic ootitis externa Allergic otitis externa Allergic pharyngitis Allergic prayingitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis Allergic renandation reaction |
| Administration site rash Administration site recall reaction Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic cosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic keratitis Allergic hepatitis Allergic hepatitis Allergic wyocarditis Allergic myocarditis Allergic oedema Allergic oetitis externa Allergic oetitis externa Allergic cotitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis Allergic sinusitis |
| Administration site recall reaction Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic keratitis Allergic hepatitis Allergic bronchitis Allergic wocarditis Allergic procarditis Allergic myocarditis Allergic oedema Allergic oetitis externa Allergic otitis externa Allergic pharyngitis Allergic prayingitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis |
| Administration site urticaria Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic cystitis Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic granulomatous angiitis Allergic hepatitis Allergic hepatitis Allergic wocarditis Allergic wocarditis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis externa Allergic pharyngitis Allergic praspiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis |
| Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic cystitis Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic hepatitis Allergic hepatitis Allergic variotis Allergic odema Allergic otitis externa Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis |
| Allergic bronchitis Allergic cough Allergic cystitis Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic hepatitis Allergic wyocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic sinusitis |
| Allergic colitis Allergic cough Allergic cystitis Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic keratitis Allergic wyocarditis Allergic oedema Allergic ootitis externa Allergic otitis externa Allergic pharyngitis Allergic pranyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic sinusitis Allergic transfusion reaction |
| Allergic cough Allergic cystitis Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic keratitis Allergic myocarditis Allergic oedema Allergic ootitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic cystitis Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic hepatitis Allergic myocarditis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic eosinophilia Allergic gastroenteritis Allergic granulomatous angiitis Allergic hepatitis Allergic keratitis Allergic wyocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic gastroenteritis Allergic pranulomatous angiitis Allergic hepatitis Allergic keratitis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic granulomatous angiitis Allergic hepatitis Allergic keratitis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic hepatitis Allergic keratitis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic keratitis Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic myocarditis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic otitis externa Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic otitis media Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic pharyngitis Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic transfusion reaction |
| Allergic respiratory symptom<br>Allergic sinusitis<br>Allergic transfusion reaction |
| Allergic sinusitis Allergic transfusion reaction |
| Allergic transfusion reaction |
| Allergy alert test positive |
| Allergy test positive |
| Allergy to immunoglobulin therapy |
| Allergy to surgical sutures |
| Allergy to vaccine |
| Alveolitis allergic |
| Anaphylactic reaction |
| Anaphylactic shock |
| Anaphylactic transfusion reaction |
| Anaphylactoid reaction |
| Anaphylactoid shock |
| Anaphylaxis treatment |

| Preferred Term |
|----------------------------------------------------------|
| Angioedema |
| Antiallergic therapy |
| Antiendomysial antibody positive |
| Anti-neutrophil cytoplasmic antibody positive vasculitis |
| Aortitis |
| Application site dermatitis |
| Application site eczema |
| Application site hypersensitivity Application site rash |
| Application site recall reaction |
| Application site urticaria |
| Application site vasculitis |
| Arteritis |
| Arteritis coronary |
| Arthritis allergic |
| Aspirin-exacerbated respiratory disease |
| Atopy |
| Behcet's syndrome |
| Blepharitis allergic |
| Blood immunoglobulin E abnormal |
| Blood immunoglobulin E increased |
| Bromoderma |
| Bronchospasm |
| Capillaritis |
| Catheter site dermatitis |
| Catheter site eczema |
| Catheter site hypersensitivity |
| Catheter site rash |
| Catheter site urticaria |
| Catheter site vasculitis |
| Cerebral arteritis |
| Chronic eosinophilic rhinosinusitis |
| Chronic hyperplastic eosinophilic sinusitis |
| Chronic pigmented purpura |
| Circulatory collapse |
| Circumoral oedema |
| Cogan's syndrome |
| Conjunctival oedema |
| Conjunctivitis allergic |
| Contact stomatitis |
| Contrast media allergy |
| Contrast media reaction |

| Preferred Term |
|-------------------------------------------------------|
| Corneal oedema |
| Cutaneous vasculitis |
| Dennie-Morgan fold |
| Dermatitis |
| Dermatitis acneiform |
| Dermatitis allergic |
| Dermatitis atopic |
| Dermatitis bullous |
| Dermatitis contact |
| Dermatitis exfoliative |
| Dermatitis exfoliative generalised |
| Dermatitis herpetiformis |
| Dermatitis infected |
| Dermatitis psoriasiform |
| Device allergy |
| Diabetic arteritis |
| Dialysis membrane reaction |
| Diffuse vasculitis |
| Distributive shock |
| Documented hypersensitivity to administered product |
| Drug cross-reactivity |
| Drug eruption |
| Drug hypersensitivity |
| Drug provocation test |
| Drug reaction with eosinophilia and systemic symptoms |
| Eczema |
| Eczema infantile |
| Eczema nummular |
| Eczema vaccinatum |
| Eczema vesicular |
| Eczema weeping |
| Encephalitis allergic |
| Encephalopathy allergic |
| Epidermal necrosis |
| Epidermolysis |
| Epidermolysis bullosa |
| Epiglottic oedema |
| Erythema induratum |
| Erythema multiforme |
| Erythema nodosum |
| Exfoliative rash |
| Eye allergy |

| Preferred Term |
|------------------------------------|
| Eye oedema |
| Eye swelling |
| Eyelid oedema |
| Face oedema |
| Fixed drug eruption |
| Giant papillary conjunctivitis |
| Gingival oedema |
| Gingival swelling |
| Gleich's syndrome |
| Granulomatosis with polyangiitis |
| Haemorrhagic urticaria |
| Haemorrhagic vasculitis |
| Hand dermatitis |
| Henoch-Schonlein purpura |
| Henoch-Schonlein purpura nephritis |
| Heparin-induced thrombocytopenia |
| Hereditary angioedema |
| Hypersensitivity |
| Hypersensitivity vasculitis |
| Idiopathic angioedema |
| Idiopathic urticaria |
| Immediate post-injection reaction |
| Immune thrombocytopenic purpura |
| Immune tolerance induction |
| Immune-mediated adverse reaction |
| Implant site dermatitis |
| Implant site hypersensitivity |
| Implant site rash |
| Implant site urticaria |
| Incision site dermatitis |
| Incision site rash |
| Infusion site dermatitis |
| Infusion site eczema |
| Infusion site hypersensitivity |
| Infusion site rash |
| Infusion site recall reaction |
| Infusion site urticaria |
| Infusion site vasculitis |
| Injection site dermatitis |
| Injection site eczema |
| Injection site hypersensitivity |
| Injection site rash |

| Preferred Term |
|---------------------------------------|
| Injection site recall reaction |
| Injection site urticaria |
| Injection site vasculitis |
| Instillation site hypersensitivity |
| Instillation site rash |
| Instillation site urticaria |
| Interstitial granulomatous dermatitis |
| Intestinal angioedema |
| lodine allergy |
| Kaposi's varicelliform eruption |
| Kawasaki's disease |
| Kounis syndrome |
| Langerhans' cell histiocytosis |
| Laryngeal oedema |
| Laryngitis allergic |
| Laryngospasm |
| Laryngotracheal oedema |
| Limbal swelling |
| Lip oedema |
| Lip swelling |
| Lupus vasculitis |
| Mast cell degranulation present |
| Medical device site dermatitis |
| Medical device site eczema |
| Medical device site hypersensitivity |
| Medical device site rash |
| Medical device site recall reaction |
| Medical device site urticaria |
| Medical device site vasculitis |
| Microscopic polyangiitis |
| Mouth swelling |
| Mucocutaneous rash |
| Multiple allergies |
| Nephritis allergic |
| Nikolsky's sign |
| Nodular rash |
| Nodular vasculitis |
| Ocular vasculitis |
| Oculomucocutaneous syndrome |
| Oculorespiratory syndrome |
| Oedema mouth |
| Oral allergy syndrome |

| Preferred Term |
|-------------------------------------------------|
| Oropharyngeal blistering |
| Oropharyngeal spasm |
| Oropharyngeal swelling |
| Palatal oedema |
| Palatal swelling |
| Palisaded neutrophilic granulomatous dermatitis |
| Palpable purpura |
| Pathergy reaction |
| Periorbital oedema |
| Pharyngeal oedema |
| Polyarteritis nodosa |
| Polymyalgia rheumatica |
| Pruritus allergic |
| Pseudovasculitis |
| Pulmonary vasculitis |
| Radiation vasculitis |
| Radioallergosorbent test positive |
| Rash |
| Rash erythematous |
| Rash follicular |
| Rash generalised |
| Rash macular |
| Rash maculo-papular |
| Rash maculovesicular |
| Rash morbilliform |
| Rash neonatal |
| Rash papulosquamous |
| Rash pruritic |
| Rash pustular |
| Rash rubelliform |
| Rash scarlatiniform |
| Rash vesicular |
| Reaction to azo-dyes |
| Reaction to colouring |
| Reaction to drug excipients |
| Reaction to preservatives |
| Red man syndrome |
| Renal arteritis |
| Renal vasculitis |
| Retinal vasculitis |
| Rheumatoid vasculitis |
| Rhinitis allergic |

| Preferred Term |
|-------------------------------------------|
| Scleral oedema |
| Scleritis allergic |
| Scrotal oedema |
| Segmented hyalinising vasculitis |
| Serum sickness |
| Serum sickness-like reaction |
| Shock |
| Shock symptom |
| Skin necrosis |
| Skin reaction |
| Skin test positive |
| Solar urticarial |
| Solvent sensitivity |
| Stevens-Johnson syndrome |
| Stoma site hypersensitivity |
| Stoma site rash |
| Swelling face |
| Swollen tongue |
| Takayasu's arteritis |
| Temporal arteritis |
| Thromboangiitis obliterans |
| Tongue oedema |
| Toxic epidermal necrolysis |
| Toxic skin eruption |
| Tracheal oedema |
| Type 2 lepra reaction |
| Type I hypersensitivity |
| Type II hypersensitivity |
| Type III immune complex mediated reaction |
| Type IV hypersensitivity reaction |
| Urticaria |
| Urticaria cholinergic |
| Urticaria chronic |
| Urticaria contact |
| Urticaria papular |
| Urticaria physical |
| Urticaria pigmentosa |
| Urticaria vesiculosa |
| Urticarial vasculitis |
| Vaccination site dermatitis |
| Vaccination site eczema |
| Vaccination site exfoliation |

| Preferred Term |
|-----------------------------------|
| Vaccination site hypersensitivity |
| Vaccination site rash |
| Vaccination site recall reaction |
| Vaccination site urticaria |
| Vaccination site vasculitis |
| Vaccination site vesicles |
| Vaginal exfoliation |
| Vaginal ulceration |
| Vascular purpura |
| Vasculitic rash |
| Vasculitis |
| Vessel puncture site rash |
| Vessel puncture site vesicles |
| Vulval ulceration |
| Vulvovaginal rash |
| Vulvovaginal ulceration |

# APPENDIX 10. AESI – SLOWING OF VENTRICULAR REPOLARIZATION

| Preferred Term |
|----------------------------------------|
| Electrocardiogram QT interval abnormal |
| Electrocardiogram QT prolonged |
| Long QT syndrome |
| Long QT syndrome congenital |
| Torsade de pointes |
| Ventricular tachycardia |

# APPENDIX 11. AESI – HEPATIC EFFECTS

| Acute hepatic failure Acute yellow liver atrophy Ascites Asterixis Bacterascites Biliary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Galbladder varices Galbladder varices Gastric variceal ligation Gastric variceal ligation Gastric varices hemorrhage Hepatic cirrhosis Hepatic circhosis Hepatic diffication Hepatic circhosis Hepatic diffication Hepatic circhosis Hepatic hepatic hyprophylaxis Hepatic hydrothorax Hepatic fibrosis Hepatic hydrothorax Hepatic necephalopathy prophylaxis Hepatic lesion Hepatic teston-fibrosis Hepatic teston-fibrosis Hepatic steato-fibrosis Hepaticular foamy cell syndrome Hepatocellular injury Hepatocellular injury | Preferred Term |
|---|---|
| Acute yellow liver atrophy Ascites Asterixis Bacterascites Biliary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal injection Gastric varices haemorrhage Hepatectomy Hepatic calcification Hepatic cirrhosis Hepatic cirrhosis Hepatic inflitration eosinophilic Hepatic hepatic inspection Hepatic inspection Hepatic inspection Hepatic encephalopathy Hepatic encephalopathy Hepatic encephalopathy Hepatic encephalopathy Hepatic inflitration eosinophilic Hepatic inspection Hepatic testoon Hepatic testoos Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatitic steato-fibrosis Hepatitic steato-fibrosis Hepatitic steato-fibrosis Hepatitic steato-fibrosis Hepatitis fulminant Hepatocellular foamy cell syndrome | Acute hepatic failure |
| Ascites Asterixis Bacterascites Biliary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatic calcification Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic infiltration eosinophilic Hepatic steatos-fibrosis Hepatic flura filary disease Hepatocellular foamy cell syndrome | Acute on chronic liver failure |
| Asterixis Bacterascites Biliary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal ligation Gastric variceal ligation Gastric varices haemorrhage Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy Hepatic encephalopathy Hepatic infiltration eosinophilic Hepatic infiltration eosinophilic Hepatic tesion Hepatic steatosis Hepatic fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic fliura disease Hepatocellular foamy cell syndrome | Acute yellow liver atrophy |
| Baltary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatectomy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic influre encephalopathy Hepatic influre hepatic fibrosis Hepatic fibrosis Hepatic inflictation eosinophilic Hepatic lesion Hepatic steato-fibrosis | Ascites |
| Biliary cirrhosis Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal ligation Gastric variceal ligation Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic fibrosis Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic seato-fibrosis Hepatic seato-fibrosis Hepatic steato-fibrosis Hepatitis fulminant Hepatocellular foamy cell syndrome | Asterixis |
| Biliary cirrhosis primary Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal ligation Gastric variceal ligation Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy Hepatic fibrosis Hepatic fibrosis Hepatic fillure Hepatic infiltration eosinophilic Hepatic steato-fibrosis | Bacterascites |
| Biliary fibrosis Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatic atrophy Hepatic atrophy Hepatic acloification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic lesion Hepatic lesion Hepatic recrosis Hepatic necrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic fulminant Hepatocellular foamy cell syndrome | Biliary cirrhosis |
| Cholestatic liver injury Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices Gastric varices Gastric varices Hepatic atrophy Hepatic atrophy Hepatic aclification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic necrosis Hepatic steato-fibrosis | Biliary cirrhosis primary |
| Chronic hepatic failure Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatic atrophy Hepatic aclification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic fibrosis Hepatic filbrosis Hepatic lesion Hepatic infiltration eosinophilic Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatit steatosis Hepatitis fulminant Hepatocellular foamy cell syndrome | Biliary fibrosis |
| Coma hepatic Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic aclification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic infiltration eosinophilic Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Cholestatic liver injury |
| Cryptogenic cirrhosis Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices haemorrhage Hepatic atrophy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic failure Hepatic filorosis Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis | Chronic hepatic failure |
| Diabetic hepatopathy Drug-induced liver injury Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices Gastric varices Gastric varices Gastric varices Hepatectomy Hepatic atrophy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy prophylaxis Hepatic failure Hepatic failure Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic lession Hepatic steato-fibrosis | Coma hepatic |
| Drug-induced liver injury Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices Gastric varices Gastric varices Gastric varices Gastric varices Hepatectomy Hepatic atrophy Hepatic alcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatit sfulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Cryptogenic cirrhosis |
| Duodenal varices Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices Gastric varices Gastric varices Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic infiltration eosinophilic Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatit steatosis Hepatitosiliary disease Hepatocellular foamy cell syndrome | Diabetic hepatopathy |
| Gallbladder varices Gastric variceal injection Gastric variceal ligation Gastric varices Gastric varices Gastric varices Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Drug-induced liver injury |
| Gastric variceal ligation Gastric varices Gastric varices Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic fibrosis Hepatic fibrosis Hepatic fibrosis Hepatic fibrosis Hepatic seasonophilic Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Duodenal varices |
| Gastric variceal ligation Gastric varices Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis | Gallbladder varices |
| Gastric varices Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic steato-fibrosis | Gastric variceal injection |
| Gastric varices haemorrhage Hepatectomy Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic failure Hepatic fibrosis Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepaticit fulminant Hepatocellular foamy cell syndrome | Gastric variceal ligation |
| Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatolliary disease Hepatocellular foamy cell syndrome | Gastric varices |
| Hepatic atrophy Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatobiliary disease Hepatocellular foamy cell syndrome | Gastric varices haemorrhage |
| Hepatic calcification Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis | Hepatectomy |
| Hepatic cirrhosis Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic atrophy |
| Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic fibrosis Hepatic steatosis Hepatic steatosis Hepatic foamy cell syndrome | Hepatic calcification |
| Hepatic encephalopathy prophylaxis Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic cirrhosis |
| Hepatic failure Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic stolminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic encephalopathy |
| Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic fibrosis Hepatic steatosis Hepatic steatosis Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic encephalopathy prophylaxis |
| Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic failure |
| Hepatic infiltration eosinophilic Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic fibrosis |
| Hepatic lesion Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic hydrothorax |
| Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic infiltration eosinophilic |
| Hepatic steato-fibrosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic lesion |
| Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic necrosis |
| Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic steato-fibrosis |
| Hepatobiliary disease Hepatocellular foamy cell syndrome | Hepatic steatosis |
| Hepatocellular foamy cell syndrome | Hepatitis fulminant |
| | Hepatobiliary disease |
| Hepatocellular injury | Hepatocellular foamy cell syndrome |
| | Hepatocellular injury |

| Preferred Term |
|--------------------------------------------|
| Hepatopulmonary syndrome |
| Hepatorenal failure |
| Hepatorenal syndrome |
| Hepatotoxicity |
| Intestinal varices |
| Intestinal varices haemorrhage |
| Liver and small intestine transplant |
| Liver dialysis |
| Liver disorder |
| Liver injury |
| Liver operation |
| Liver transplant |
| Lupoid hepatic cirrhosis |
| Minimal hepatic encephalopathy |
| Mixed liver injury |
| Nodular regenerative hyperplasia |
| Non-alcoholic fatty liver |
| Non-alcoholic steatohepatitis |
| Non-cirrhotic portal hypertension |
| Oedema due to hepatic disease |
| Oesophageal varices haemorrhage |
| Peripancreatic varices |
| Portal fibrosis |
| Portal hypertension |
| Portal hypertensive enteropathy |
| Portal hypertensive gastropathy |
| Portal vein cavernous transformation |
| Portal vein dilatation |
| Portopulmonary hypertension |
| Renal and liver transplant |
| Retrograde portal vein flow |
| Reye's syndrome |
| Reynold's syndrome |
| Splenic varices |
| Splenic varices haemorrhage |
| Steatohepatitis |
| Subacute hepatic failure |
| Varices oesophageal |
| Varicose veins of abdominal wall |
| Anorectal varices |
| Anorectal varices haemorrhage |
| Intrahepatic portal hepatic venous fistula |

| Preferred Term |
|-----------------------------------------------------|
| Peritoneovenous shunt |
| Portal shunt |
| Portal shunt procedure |
| Small-for-size liver syndrome |
| Spider naevus |
| Splenorenal shunt |
| Splenorenal shunt procedure |
| Spontaneous intrahepatic portosystemic venous shunt |
| Stomal varices |

### **APPENDIX 12. AESI – SEXUAL DYSFUNCTION**

| Anorgasmia |
|--------------------------------|
| Disturbance in sexual arousal |
| Dyspareunia |
| Ejaculation delayed |
| Ejaculation disorder |
| Ejaculation dysfunction |
| Ejaculation failure |
| Erectile dysfunction |
| Female orgasmic disorder |
| Female sexual arousal disorder |
| Female sexual dysfunction |
| Inadequate lubrication |
| Libido decreased |
| Libido disorder |
| Loss of libido |
| Male orgasmic disorder |
| Male sexual arousal disorder |
| Male sexual dysfunction |
| Orgasm abnormal |
| Orgasmic sensation decreased |
| Sexual dysfunction |
| Vulvovaginal dryness |